CLINICAL TRIAL: NCT00836797
Title: Phase I Radiographic Assessment of Bone Regeneration in Alveolar Sockets With PLGA Bioscaffold After Teeth Extraction
Brief Title: Radiographic Assessment of Bone Regeneration in Alveolar Sockets With PLGA Scaffold
Status: Completed | Type: Observational
Sponsor: Bio-Scaffold International Pte Ltd (Industry)
Collaborators: National University Hospital, Singapore (Other); Saveetha University (Other)
Responsible Party: Dr. Victor Tai Weng Fan/ Assistant Professor, Faculty of Dentistry, National University of Singapore
Other Study IDs: BSI-001-VF; DSRB A/06/404
Record Dates: First submitted 2009-02-03; First posted 2009-02-04 (Estimated); Last update posted 2009-02-04 (Estimated); Status verified 2009-02

CONDITIONS: Preservation of Alveolar Bone Height With PLGA Bioscaffold
Keywords: Alveolar Bone Loss; Alveolar ridge; Alveolar Process
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1 Case with scaffold: This group of patients will be having a placement of PLGA bioscaffold in the alveolar socket after teeth extraction
- 2 Control without scaffold: The Alveolar socket will be left to heal and no treatment/scaffold placement will be done

SUMMARY:
After extraction of a tooth, the bony socket heals naturally but due to the absent of the tooth and any presence of support in the socket, bone resorption occur both vertically and bucco lingually or bucco palataly. This bony resorption ultimately effects a lot of things like - the support for the adjacent teeth become weak, the shallow ridge makes it difficult for future prosthesis retention, and less bony support for any implant placement in the future which is the most popular and effective way of tooth replacement now a days. So now a days keeping the integrity and contour of the alveolar bony socket is very important for the patients future rehabilitation. The use of scaffold will help to maintain the integrity of the alveolar bony socket thus provides a vital support for the adjacent teeth, preserve the alveolar crest height, maintain the bony contour, helps to prevent bleeding, and most importantly it will help in bone regeneration which is the vital factor for future rehabilitation.

DETAILED DESCRIPTION:
A case controlled study design is adopted. Patients who will be having extraction of any tooth including surgical extraction but not due to any periodontal reasons are selected. Consent of the patient will be taken for the procedure and all the effects and possibilities will be explained to the patients. Extraction will be done and scaffold material will be placed inside the socket. Sockets with the scaffold will be the variable studied and the sockets without scaffold placed inside the sockets will be the control group. An OPG x ray will be taken with the head position standardized by a positioning device. A second x-ray will be taken following the same technique after two months (for assessment of bone healing as is practiced normally) and a final x-ray will be taken after 3 months of the first x-ray (normally done in clinics for assessment of socket prior to implantation.

The OPG x ray is taken with the patient biting on a bite plate device fabricated with an embedded wire inside which is radiopague. If the distance from the wire line (the occlusal plane) to the alveolar bony height is 'a' and if the actual diameter of the metallic ball is 'b' and radiographic ball diameter is 'c' then the equation ( a×b)/c will give us the distance of the alveolar bony crest from the wire line. The measurements taken will determine if the distance of the alveolar crest from the wire line remained the same or has increased. If it remains the same, it will suggest that the scaffold material had maintained the socket and prevented alveolar bone resorption, but if the distance increases that will indicate vertical loss of alveolar bone and the extent measured can be compared with sockets without the support of an immediate post-extraction scaffold. This study will determine firstly whether the scaffold allows for bone regeneration in human alveolar sockets in the normal time and secondly whether it would help to preserve alveolar bone height as compared to cases without scaffold.

Consent of the selected patient will be taken for the procedure. Extraction will be done and scaffold material will be placed inside the socket. Socket with the scaffold will be our cases and the socket without scaffold will be the control group in multiple extraction cases. Radiographic assessment will be done to assess bone regeneration at the prescribed pre-extraction stage, at the 2 months bone healing stage and at the 3 months (from initial extraction) implant planning stage as in usual clinical practice . Assessment of the bony height is made with the prescribed formula from the radiographs taken and comparison will be made with the control cases. The following are the criteria for selecting the patients.

ELIGIBILITY:
Inclusion Criteria:

1. Under going extraction of tooth including the surgical extraction.
2. Healthy individual with no known medical problems.
3. Not allergic to foreign body.
4. Extractions which are not due to periodontal causes.

Exclusion Criteria:

1. Bony disease.
2. Bleeding disorder.
3. Allergic to foreign body.
4. Mentally retarded persons.
5. Diabetic patient.
6. Drug addict.
7. Extraction due to periodontal disease.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Dental clinic patients undergoing teeth extraction
Sampling Method: Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2007-05; Primary Completion 2007-09 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Preservation of Alveolar height | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Tai Weng Fan Victor, BDS FDSRCS, Principal Investigator — National University of Singapore, Faculty of Dentistry
Locations (2):
- Saveetha Dental College, Saveetha University, Chennai, Tamil Nadu, India
- Dental Centre, National University Hospital,, Singapore, Singapore